CLINICAL TRIAL: NCT04828564
Title: An Open-Label, Multicenter, Parallel-Group, Randomized, Phase II/III Study to Evaluate the Efficacy and Safety of Favipiravir and Ribavirin Formulation for Treatment of COVID-19
Brief Title: Efficacy and Safety of Favipiravir and Ribavirin Formulation for Treatment of COVID-19
Acronym: COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Scientific and Technological Research Council of Turkey (Other)
Collaborators: Ankara City Hospital Bilkent (Other); Istanbul Umraniye Training and Research Hospital (Unknown); Koç University (Other); Monitor CRO (Industry)
Responsible Party: Principal Investigator, Alpay Azap, Prof., MD., Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MON775.159.4
Record Dates: First submitted 2021-04-01; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: SARS-CoV2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ribavirin; favipiravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ribavirin Arm (Experimental): Ribavirin dosage: 200 mg oral ribavirin capsules for 5 days
  Regimen: 1200 mg loading dose on day-1 (three capsules in the morning and three capsules in the evening) followed by 800 mg/day maintenance dose (two capsules in the morning and two capsules in the evening) on day-2 to day-5.
  Interventions: Drug: Ribavirin Capsules
- Favipiravir Arm (Active Comparator): Favipiravir dosage: 200 mg oral favipiravir tablets for 5 days
  Regimen: 2x1600 mg loading dose on day-1 (eight tablets in the morning and eight tablets in the evening) followed by 2x600 mg maintenance dose (three tablets in the morning and three tablets in the evening) on day-2 to day-5.
  Interventions: Drug: Favipiravir

INTERVENTIONS:
Drug: Ribavirin Capsules — Ribavirin 200 mg capsules
  Arms: Ribavirin Arm
Drug: Favipiravir — Favipiravir 200 mg tablets
  Arms: Favipiravir Arm

SUMMARY:
This is a national, multicenter, open-label, randomized, phase II/III trial that evaluates the efficacy and safety of favipiravir and ribavirin in the treatment of patients with confirmed COVID-19 observed within 72 hours. Approximately 100 patients will be randomized in 1:1 ratio and divided into two groups.

DETAILED DESCRIPTION:
The clinical picture of COVID-19 disease is in a broad spectrum, which includes asymptomatic infection, a mild upper respiratory tract infection, respiratory failure, and even severe viral pneumonia with death. The alarming levels of spread and severity of COVID-19 caused a global emergency and this outbreak has been characterized as a pandemic by the World Health Organization (WHO).

Coronavirus entry into host cells is an important determinant of viral infectivity and pathogenesis. SARS-CoV S1 contains a receptor-binding domain (RBD) that specifically recognizes angiotensin-converting enzyme 2 (ACE2) as its receptor. SARS-CoV spike needs to be proteolytically activated at the S1/S2 boundary, such that S1 dissociates and S2 undergoes a dramatic structural change. These SARS-CoV entry-activating proteases include cell surface protease TMPRSS2 and lysosomal proteases cathepsins. These features of SARS-CoV entry contribute to its rapid spread and severe symptoms and high fatality rates of infected patients.

Ribavirin is a guanosine analog that interferes with the replication of RNA and DNA viruses. Ribavirin was used during the Severe Acute Respiratory Syndrome (SARS) outbreak in combination with corticosteroids, which have an anti-inflammatory effect. Favipiravir is a substrate for viral RNA-dependent RNA polymerase (RdRp) and showed anti-influenza virus activity. Favipiravir is effective against other RNA viruses, poliovirus, rhinovirus, and respiratory syncytial virus and evaluated and developed as a broad spectrum anti-RNA virus drug, including lethal RNA virus infections.

According to national guidelines, Favipiravir treatment is applied to COVID-19 infection in Turkey. The main purpose of this study is to obtain efficacy and safety data for ribavirin and favipiravir in the Turkish patient cohort diagnosed with COVID-19.

This study designed as an open-label, multicenter, parallel-group, randomized, phase II/III clinical drug trial.

This study will be conducted in 4 sites.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients aged 18 years and older infected with the SARS-CoV-2 virus.
* Patients that have COVID-19 symptoms within 72 hours and have a positive PCR test result.
* Patients in a stable clinical condition and referred as outpatient for COVID-19 infection.
* Patients who sign the informed consent before the any study procedures.

Exclusion Criteria:

* Patients who have required hospitalization.
* Patients who have required intensive care.
* Patients who do not sign the informed consent.
* Any condition that in the investigator's judgement might interfere with study procedures or the ability of the patient to adhere to and complete the study.
* Patients who have been participating in any other clinical trial.
* Severe liver failure (Child Pugh score ≥ C, transaminase>5 times the upper limit of normal (ULN).
* Severe renal failure (GFR ≤30 mL/min/1.73 m2) or continuous dialysis (hemodialysis, peritoneal dialysis) or continuous renal replacement therapy.
* Severe cardiac disease.
* History of hypersensitivity to either ribavirin/favipiravir.
* Pregnant or breast-feeding.
* Patients who cannot use appropriate contraceptive method during and after the study.
* Patients who are treated with any other treatment agent for COVID-19 in the last 90 days.
* Patients who had COVID-19 vaccination.
* Patients who had ribavirin/favipiravir for any reason in the past 72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospitalized patient rates | 15 days
  The number of hospitalized patients

SECONDARY OUTCOMES:
Mortality rate | 15 days
  All-cause mortality rate
Time from randomization to relief of symptoms | 15 days
  The duration (days) from start of treatment to relief of clinical symptoms
Viral clearance | 15 days
  The day of viral clearance evaluated by real-time polymerase chain reaction (RT-PCR)
Changes in angiotensin-converting enzyme 2 (ACE2) receptor levels | 15 days
  Detection of RNA and/or protein levels of ACE2 gene in plasma samples via quantitative RT-PCR and/or flow cytometry
Changes in transmembrane protease serine II (TMPRSS2) activity | 15 days
  Assessment of proteolytic activity of TMPRSS2
Emergency room visit rates of patients | 15 days
  The number of emergency room visits of patients (not hospitalized)
Time to emergency room visit | 15 days
  The time (days) until the emergency room visit
Time to hospitalization | 15 days
  The time (days) until the hospitalization
Inpatient length of stay | 15 days
  Length of stay in the hospital (days)
Time to ICU admission | 15 days
  The time (days) until admission to intensive care unit
Time to intubation | 15 days
  The time (days) until intubation
Family members rates with PCR positive test results | 15 days
  The number of family members with PCR positive
Changes in vital signs from baseline | 15 days
  Clinical evaluation of systolic and diastolic blood pressure, pulse, respiratory rate, fever, oxygen saturation changes from baseline until the end of study
Number/characteristics of AEs and SAEs | 28 days
  Number/characteristics of Adverse Event (AE) and Serious Adverse Event (SAE) related to study drug or hematological and biochemical parameters from baseline until the end of study

CONTACTS AND LOCATIONS:
Locations (4):
- Turkey (Türkiye) (4):
  - Ankara University, School of Medicine, Ankara, Cebeci
  - Ankara City Hospital, Ankara
  - Koc University Hospital, Istanbul
  - Umraniye Training and Research Hospital, Istanbul